CLINICAL TRIAL: NCT06010069
Title: The Relationship Between the Frequency of Intraoperative Hypothermia and Fragility Scores in the Elderly Patient Group. Prospective Cohort Study
Brief Title: The Relationship Between the Frequency of Intraoperative Hypothermia and Fragility Scores
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Fatma Nur Arslan, Medical Docdor, Kirsehir Ahi Evran Universitesi
Other Study IDs: 22.11.2022 No: 2022-21/187
Record Dates: First submitted 2023-08-21; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Hypothermia; Anesthesia; Fragility
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- pre-frail patients: That patient group have clinical frailty scale scores 1,2 or 3 which is accepted as non-frail.
  Interventions: Diagnostic Test: body temperature measurament
- frail patients: That patient group have clinical frailty scale scores 4 or 5 which is accepted as frail.
  Interventions: Diagnostic Test: body temperature measurament
- very frail patients: That patient group have clinical frailty scale scores 6,7,8 or 9 which is accepted as severly frail.
  Interventions: Diagnostic Test: body temperature measurament

INTERVENTIONS:
Diagnostic Test: body temperature measurament — body temperature of every patient was measured with tympanic thermometer during surgical procedure

SUMMARY:
The goal of this observational study is to compare frequency of intraoperative hypothermia between fragilitly groups of eldery patients who underwent orthopedic surgical procedures.

It aims to answer those questions:

* İs there any difference between fragility groups in terms of hypothermia frequency during orthopedic surgical procedures?
* Are there any other factors that influence the frequency of hypothermia such as age, body mass index, room temperature etc. ? Participants body temperature before anestesia application,and before surgery had started was measured and measurament was done during whole procedure. Measuraments had been done by tympanic thermometer.

ELIGIBILITY:
Inclusion Criteria:

* Elective Orthopedic Surgery Candidates
* 65 years old or older

Exclusion Criteria:

* Emergency surgery
* Patiens who required multiple (2 or more) blood component transfusions
* Neurologic disorders
* tyroid dysfunction
* Patiens who are already hypothermic before surgery

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Our candidates was choosen from patiens who scheduled for elective orthopedic surgeries in Kirsehir education and research hospital. We have enrolled patients who accepted to be a partician for this study after obtaining their informed consent. Elective Orthopedic Surgery. All of our participants were 65 years old or older.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
frequency of hypothermia | during the orthopedic surgical procedure
  difference between frailty groups in terms of frequency of hypothermia

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Eğitim ve Araştırma Hastanesi, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
After the statistical analyzes we will most likely to share IPDs